CLINICAL TRIAL: NCT02344563
Title: A Randomized, Single-dose, Two-way Crossover Study to Evaluate Bioequivalence of Two Formulations of Meropenem In Healthy Volunteers(Meropenem Intravenous Injection) After Intravenous Infusion
Brief Title: Bioequivalence of Two Formulations of Meropenem Intravenous Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: YSP-RBH3012-03
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: volunteers

ARMS (2):
- Meropem (Experimental): 0.5g/vial,one vial
  Interventions: Drug: Meropem; Drug: Mepem
- Mepem (Active Comparator): 0.25g/vial ,two vials
  Interventions: Drug: Meropem; Drug: Mepem

INTERVENTIONS:
Drug: Meropem
Drug: Mepem

SUMMARY:
A randomized, single-dose, two-way crossover study to evaluate bioequivalence of two formulations of meropenem (meropenem intravenous injection 0.5 g) after intravenous infusion in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subjects between 20-45 years of age.
* Body weight within 80-120% of ideal body weight and higher than or equal to 50 kg for male subjects and 45 kg for female subjects.

  * Ideal body weight (kg) = [height (cm) - 80] × 0.7 for male subjects
  * Ideal body weight (kg) = [height (cm) - 70] × 0.6 for female subjects
* Acceptable medical history and physical examination including:

no particular clinically significant abnormality in X-ray and ECG results within six months prior to study. no particular clinical significance in general disease history within two months prior to study.

* Acceptable vital signs (within normal limits or considered by the investigator or physician to be of no clinical significance) at screening, which includes pulse rate, blood pressure and body temperature.
* Acceptable clinical chemistry determinations (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study, which includes AST (SGOT), ALT (SGPT), γ-GT, alkaline phosphatase, total bilirubin, albumin, glucose, BUN, uric acid, creatinine, total cholesterol and triglyceride (TG).
* Acceptable hematology (within normal range or considered by the investigator or physician to be of no clinical significance) within two months prior to study, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials and platelets.
* Acceptable urinalysis (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study, which includes pH, blood, glucose, ketones, bilirubin and protein.
* Female subjects of childbearing potential practicing an acceptable method of birth control from at least seven days prior to study until the end of study as judged by the investigator(s) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy performed on the subject).
* Have signed the written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the clinical investigator).
* A clinically significant illness or surgery within four weeks prior to study (as determined by the investigator).
* History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years.
* History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant.
* Known or suspected history of drug abuse within lifetime as judged by the investigator.
* History of alcohol addiction or abuse within last five years as judged by the investigator.
* Have a personal history or family history of drug allergy.
* Subjects demonstrating a positive meropenem skin test screen prior to the study.
* Evidence of chronic or acute infectious diseases.
* Female subjects demonstrating a positive urine pregnancy screen prior to study.
* Female subjects who are currently breastfeeding.
* Taking any drug known to induce or inhibit hepatic drug metabolism within four weeks prior to study. Examples of inducers include: piperidines, carbamazepine, dexamethasone and rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatin, methadone and ranitidine.
* Taking any prescription medications within four weeks or any nonprescription medications (excluding flu vaccination) within two weeks prior to study.
* Use of any investigational drug within four weeks prior to study.
* Donating more than 250 mL of blood within two months prior to study or donating plasma (e.g. plasmapheresis) within two weeks prior to study.
* Any other medical reason as determined by the clinical investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adverse events and incidences | predose to 6 hours post dose

SECONDARY OUTCOMES:
Pharmacokinetic parameters | pre dose to 6 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Yuan Shi, M.D., Principal Investigator — zyshi@vghtc.gov.tw